CLINICAL TRIAL: NCT01291342
Title: Detection and Identification of Preeclampsia Via Volatile Biomarkers
Acronym: DIP
Status: Completed | Type: Observational
Sponsor: The Nazareth Hospital, Israel (Other)
Collaborators: Technion, Israel Institute of Technology (Other); HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Marwan Hakim, DoCTOR, The Nazareth Hospital, Israel
Other Study IDs: 1702
Record Dates: First submitted 2011-02-05; First posted 2011-02-08 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy; Death of Fetus, Early Pregnancy; Uremia in Pregnancy Without Hypertension
Keywords: Pregnancy; Preeclampsia; Volatile biomarkers; Chemical sensors; Nanomaterials; Nanosensors; NA-NOSE
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Preeclampsia: 30 preeclamptic pregnant women with gestational age >24 weeks and no chronic medical disorders who are not in labor and their fetus is alive.
- Normal pregnancy: 30 normotensive pregnant women with gestational age >24 weeks and no chronic medical disorders who has no obstetrical problems, not in labor and their fetus is alive.
- Healthy non-pregnant: 30 healthy non-pregnant control women not on medications and has not delivered a baby or conceived during the year before the breath collection

SUMMARY:
Preeclampsia is a form of hypertension that is unique to human pregnancy. The incidence of the disease ranges between 2 and 7 percent in healthy nulliparous women. The etiology of preeclampsia is unknown.

Women with preeclampsia may exhibit a symptom complex ranging from minimal BP elevation to derangements of multiple organ systems. The renal, hematologic, and hepatic systems are most likely to be involved.

More than 100 clinical, biophysical, and biochemical tests have been recommended to predict or identify the patient at risk for the future development of the disease.

The results of the pooled data for the various tests and the lack of agreement between serial tests suggest that none of these clinical tests is sufficiently reliable for use as a screening test in clinical practice. As a result there is obviously a great need to develop a novel technology for the early detection of this pregnancy complication before its clinical manifestations appear. An early detection can help in early treatment to prevent or at least minimize the sequel of this disease.

The aim of this project is the early detection of "Preeclampsia" and other pregnancy complications using volatile biomarkers appearing in exhaled breath and/or blood samples, using a simple and inexpensive toll termed NA-NOSE.

Phase-I: The primary phase of this project is the comparison between volatile biomarkers' patterns of pregnant women suffering from "Preeclampsia", pregnant women that are considered to have "Normal Pregnancy", and healthy "Non-Pregnant" women.

Phase-II: The secondary phase of this project is the ability to predict "Preeclampsia", as compared, head-to-head, with other potential predictors used in the current clinical practice.

DETAILED DESCRIPTION:
Preeclampsia is a form of hypertension that is unique to human pregnancy. The clinical findings of preeclampsia can manifest as either a maternal syndrome (hypertension and proteinuria with or without other multisystem abnormalities) or as a fetal syndrome (fetal growth restriction, reduced amniotic fluid, and abnormal oxygenation).

The incidence of preeclampsia ranges between 2 and 7 percent in healthy nulliparous women. In these women, preeclampsia is generally mild, with the onset near term or intrapartum (75 percent of cases), and the condition conveys only a minimally increased risk for adverse pregnancy outcome. In contrast, the incidence and severity of preeclampsia are substantially higher in women with multifetal gestation, chronic hypertension, previous preeclampsia, pregestational diabetes mellitus, and in those with preexisting thrombophilias.

The etiology of preeclampsia is unknown. Many theories have been suggested, but most of them have not withstood the test of time. Some of these theories: Abnormal trophoblast invasion, coagulation abnormalities, vascular endothelial damage, cardiovascular maladaptation, immunologic phenomena, genetic predisposition and dietary deficiencies or excesses.

Preeclampsia is a clinical syndrome that embraces a wide spectrum of signs and symptoms that have been clinically observed to develop alone or in combination. The classic triad of preeclampsia includes: hypertension, proteinuria, and edema. However, there is now universal agreement that edema should not be considered as part of the diagnosis of preeclampsia. The diagnosis of preeclampsia requires the presence of an elevated blood pressure (BP) with proteinuria,3 usually starting after the 20th week of the pregnancy, but the severity of the disease process is generally based on the maternal BP which is considered as the traditional hallmark for diagnosis of the disease.

Women with preeclampsia may exhibit a symptom complex ranging from minimal BP elevation to derangements of multiple organ systems. The renal, hematologic, and hepatic systems are most likely to be involved.

Renal function is usually impaired in almost every case as proteinuria is always found. In preeclampsia, vasospasm and glomerular capillary endothelial swelling (glomerular endotheliosis) lead to an average reduction in GFR (glomerular filtration rate) of 25 percent below the rate for normal pregnancy. Serum creatinine is rarely elevated in preeclampsia, but uric acid is commonly increased. Despite the fact that uric acid levels are elevated in women with preeclampsia, this test is not sensitive or specific for the diagnosis of the disease.

The liver is not primarily involved in preeclampsia, and hepatic involvement is observed in only 10 percent of women with severe preeclampsia. Fibrin deposition has been found along the walls of hepatic sinusoids in preeclamptic patients with no laboratory or histologic evidence of liver involvement. When liver dysfunction does occur in preeclampsia, mild elevation of serum transaminase is most common. Bilirubin is rarely increased in preeclampsia, but when elevated, the indirect fraction predominates. Elevated liver enzymes are part of the of HELLP syndrome, a variant of severe preeclampsia.

Thrombocytopenia is the most common hematologic abnormality in women with preeclampsia. It is correlated with the severity of the disease process and the presence or absence of placental abruption. A platelet count of less than 150,000/mm3 has been reported in 32 to 50 percent of women with severe preeclampsia, And in 15 percent of cases of women with hypertension during pregnancy.

Review of the literature reveals that more than 100 clinical, biophysical, and biochemical tests have been recommended to predict or identify the patient at risk for the future development of the disease.

The results of the pooled data for the various tests and the lack of agreement between serial tests suggest that none of these clinical tests is sufficiently reliable for use as a screening test in clinical practice. As a result there is obviously a great need to develop a novel technology for the early detection of this pregnancy complication before its clinical manifestations appear. An early detection can help in early treatment to prevent or at least minimize the sequel of this disease.

Volatile Biomarkers of Preeclampsia:

The intensity of oxidative stress in women having normal pregnancy, preeclampsia, and nonpregnant women, as expressed by volatile biomarkers through exhaled breath, was studied by GC-Chromatography/Mass-Spectrometry (GC-MS)by the group of Moretti and Phillips. A 3-D display of abundance of C4-C20 alkanes and monomethylated alkanes showed that the mean volume under curve was significantly higher in preeclampsia patients than in normal pregnant women (P<003) and nonpregnant control subjects (P<005). A predictive model employing five volatile biomarkers (undecane, 6-methyltridecane, 2-methylpentane, 5-methyltetradecane, and 2-methylnonane) distinguished preeclampsia from uncomplicated pregnancy (sensitivity=92.3%, specificity=89.7%; cross-validated sensitivity=88.5%, specificity=79.3%). While promising, the clinical value of this breath test as a predictor of preeclampsia is still unknown. This could be attributed to the fact that the study focused only on the oxidative stress relation to the preeclampsia at the time metabolic pathways cannot be ignored.

A support for the latter comes from the involvement of many disorders (e.g., renal, hematologic, and hepatic), which has been found to emit volatile biomarkers, during the preeclampsia.

Putting this preliminary study into wider perspective, longitudinal studies are required to determine if increased breath biomarkers of oxidative stress, and, also, metabolic pathways during earlier stages of pregnancy can predict the onset of preeclampsia. While part of the required knowledge could be gained by means of mass-spectrometry techniques, the use of these techniques are impeded by the need for expensive equipment, the high levels of expertise required to operate such instruments, the speed required for sampling and analysis, and the need for preconcentration techniques (a technique that allows detecting only part (15-20%) of the volatile biomarkers found in the real exhaled breath).

For preeclampsia's volatile biomarker testing to become a clinical reality, several advances in the knowledge of specific preeclampsia volatile biomarkers and sensor development need to occur. Chemical sensor matrices, based on nanomaterials, are more likely to become a clinical and laboratory diagnostic tool, because they are significantly smaller, easier-to-use, and less expensive. An ideal chemical sensor for volatile biomarker analysis should be sensitive at very low analyte concentrations in the presence of water vapour (as breath samples contain 80-90% RH). Furthermore, it should respond rapidly and differently to small changes in concentration, and provide a consistent output that is specific to a given exposure.

Objectives:

The aim of this project is the early detection of "Preeclampsia" and other pregnancy complications using volatile biomarkers appearing in exhaled breath and/or blood samples, using a simple and inexpensive toll termed NA-NOSE.

Phase-I: The primary phase of this project is the comparison between volatile biomarkers' patterns of pregnant women suffering from "Preeclampsia", pregnant women that are considered to have "Normal Pregnancy", and healthy "Non-Pregnant" women.

Phase-II: The secondary phase of this project is the ability to predict "Preeclampsia", as compared, head-to-head, with other potential predictors used in the current clinical practice.

Methodology:

Study Design and Outline:

Phase-I of this study will concentrate on a cross sectional breath tests of three groups of young women who agreed to participate and signed an informed consent form that was approved by the institutional Helsinki committee in the Nazareth Hospital.

Groups:

* Preeclampsia: 30 preeclamptic pregnant women with gestational age >24 weeks and no chronic medical disorders who are not in labor and their fetus is alive. Preeclampsia is defined as blood pressure of >140/90 mm Hg on 2 separate occasions at least 4 hours but not more than one week apart with proteinuria. Proteinuria is defined as a urinary dipstick value >1+ (30mg/dL), or a 24 hour urine collection with a protein excretion of >300mg.
* Uncomplicated pregnancy: 30 normotensive pregnant women with gestational age >24 weeks and no chronic medical disorders who has no obstetrical problems, not in labor and their fetus is alive.
* Healthy controls: 30 healthy non-pregnant control women recruited mainly from employees of the Nazareth Hospital who are healthy, not on medications and has not delivered a baby or conceived during the year before the breath collection.

Breath Test Sampling for the NA-NOSE as well as the blood samples will be done in the Technion.

Chemical analysis:

The LNBD group (Technion) will determine the most pronounced electrical features for each organically functionalized nanosensor in response to the volatile biomarkers (of both breath and blood samples), and of the entire sensor array, using classical multi-linear regression models and neural network models. Different linear and nonlinear algorithms will be sought based on principal component analysis and chaotic parameters in order to reduce the dimensions of the data, and to extract the most important information. The exhaled air will also be analyzed by Gas-Chromatography/Mass-Spectrometry (GC-MS) in conjugation with thermal desorption for determining the nature and composition of the volatile biomarkers in the related breath and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* All participants are nonsmokers, non obese, young women between 18 and 40 years old who'll be able to provide breath samples.

Exclusion Criteria:

* Women taking medicines or antioxidants are excluded except the pregnant women who are on traditional prenatal vitamins and those in the preeclampsia group on antihypertensive medication.
* Obese women or those with chronic diseases and those with a history of chronic hypertension, insulin-dependent diabetes or renal disease are excluded.
* minors and insane

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women treated in the Nazareth Hospital and Emek Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Volatile Biomarkers | Volatile Biomarkers will be collected from pregnant women and analysed afterward

CONTACTS AND LOCATIONS:
Overall Officials: Marwan M Hakim, M.D, D.Sc, Principal Investigator — he Nazareth Hospital E.M.M.S
Locations (1):
- Nazareth Hospital, Nazareth, Israel